CLINICAL TRIAL: NCT04118959
Title: The Value of Atosiban on the Day of Embryo Transfer in Patients With Recurrent Implantation Failure
Brief Title: Role of Atosiban in Recurrent Implantation Failure
Acronym: RIF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al Baraka Fertility Hospital (Other)
Responsible Party: Principal Investigator, Dr. Kamal Rageh, doctor , medical director, Al Baraka Fertility Hospital
Other Study IDs: K.Rageh
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Recurrent Implantation Failure
Keywords: Recurrent implantation failure; IVF; Atosiban; Embryo Transfer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ET is the final stage of IVF which independently influences the treatment outcome. Successful embryo implantation is dependent on uterine receptivity. Atosiban is a novel class of drug which is effective in priming the uterus for implantation. It reduces uterine contractions and increases endomyometrial perfusion, both of which have potential benefits regarding improved IRs, CPR, and ongoing pregnancy rates. Atosiban has a good embryonic safety profile. It has no systemic toxicity, no mutagenic effects, and no carcinogenic effects

DETAILED DESCRIPTION:
ET is a critical step of an IVF cycle that merits the utmost attention. Its success depends on the frequency of uterine contractions, the endometrial receptivity and the quality of embryos transferred.

Uterine contractions are the most fundamental constituents of the uterine receptivity. Excessive contractions may decrease the implantation potential of embryos by expelling the embryos from the uterus. Studies have revealed a six-fold increase in uterine contractility in IVF cycles when measured before ET as compared to the condition before ovulation in natural cycles. Excessive manipulation of the cervix such as the use of tenaculum during difficult ET can also trigger uterine contractions, consequently leading to failure of embryo implantation.

IVF success rates have been potentially improved by the use of drugs that inhibit pronounced uterine contractions at the time of ET. Treatment strategies such as the use of beta-agonists or nonsteroidal anti-inflammatory agents for tocolysis have not been beneficial in IVF-ET procedures.

Atosiban is a combined oxytocin/vasopressin V1A antagonist. It functions mainly by blocking oxytocin and vasopressin V1a receptors to decrease the frequency and amplitude of uterine contractions, which enhances implantation and pregnancy rates. RIF remains unexplained in most cases, which results in considerable variation in how RIF is treated and managed. Atosiban competes with oxytocin at oxytocin receptors in endometrial cells and inhibits oxytocin-induced PGF2α release, thus inhibiting uterine contractions and increasing chances of embryo implantation and may add value in improving the outcome in RIF patients.

Recently published studies showed that atosiban inhibits oxytocin-induced PGF2α and uterine contractility, consequently leading to improved IRs. Studies have shown a considerable reduction in the frequency of uterine contractions before and after the administration of atosiban in women undergoing ET.

ELIGIBILITY:
Inclusion Criteria:

1. Women 22-40 years age
2. Body mass index- 18.5-30 kg/m 2
3. The normal uterine cavity on ultrasound scan
4. At least one good quality embryo present for transfer
5. Endometrium thickness ≥7.5 mm with endometrial volume 2-2.5 ml and good endometrial and subendometrial vascularity.

Exclusion Criteria:

* 1. Women ≥ 40 years age 2. Uterine abnormalities that can compromise the IRs (e.g., endometrial polyp, fibroids, hydrosalpinx, and adenomyosis) 3. Patients at risk of ovarian hyperstimulation syndrome 4. Patients with a history of hypersensitivity to atosiban 5. Endocrine dysfunction 6. Major organ dysfunction such as liver or kidney failure.

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: those patients with a history of recurrent implantation failure
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-11-25 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 2 weeks
  B- HCG
clinical pregnancy rate | 4 weeks
  positive fetal heart beats

CONTACTS AND LOCATIONS:
Locations (1):
- Al-BARAKA FERTILITY HOSPITAL, Adliya, Manama, Bahrain